CLINICAL TRIAL: NCT03917862
Title: The Hemostatic Potential of TDM-621 on Ascending Aortic Surgery
Brief Title: Strategy for Aortic Surgery Hemostasis
Acronym: SASH
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: 3-D Matrix UK Ltd. (Industry); InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Ricardo Ribeiro Dias, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93960818.9.1001.0068
Record Dates: First submitted 2019-02-05; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ascending Aorta Abnormality; Ascending Aortic Dissection; Ascending Aorta Aneurysm
Keywords: Ascending Aortic Surgery; Hemostasis; Ascending Aortic Dissection; Ascending Aorta Aneurysm; Bleeding
MeSH Terms: conditions — Dissection, Ascending Aorta; Aneurysm, Ascending Aorta; Hemorrhage | interventions — acetyl-(arginyl-alanyl-aspartyl-alanyl)4-amide

STUDY DESIGN:
Intervention Model Description: SASH Trial is a multicenter, prospective, open and randomized 1:1 study. Will be included 200 consecutive patients randomized to receive TDM-621 or regular procedure. It will be performed in 5 different centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group include patients which will be undergone to conventional ascending aortic surgery, according to stablished techniques.
- TDM-621 (Active Comparator): This group include patients which will be undergone to conventional ascending aortic surgery, according to stablished techniques and will receive the TDM-621 for complementary hemostasis.
  Interventions: Combination Product: TDM-621

INTERVENTIONS:
Combination Product: TDM-621 — The TDM-621 is a topic hemostatic product which will be used during ascending aortic surgery.
  Other Names: PuraStat®
  Arms: TDM-621

SUMMARY:
SASH Trial is a multicenter, prospective, open and randomized 1:1 study. The aim of this study is to evaluate the efficacy of TDM-621(Three-D Matrix- 621) (PuraStat®) on hemostasis of ascending aortic surgery. The TDM-621 is a topic hemostatic product. When in contact with blood it allowed to cover the sutures improving the hemostasis. The hypothesis is that the use of TDM-621 may reduce bleeding and the need for blood transfusion of patients undergoing ascending aortic surgeries. It will include 200 consecutive patients randomized to receive TDM-621 or regular procedure, performed in 5 different centers.

DETAILED DESCRIPTION:
According to data from the National Center for Health Statistics 2013, more than 51 million surgical procedures with hospitalized patients are conducted annually in the United States. During and postoperative bleeding is a concern for increasing the morbidity and mortality of the procedures, in addition to being sometimes associated with the need for reoperation.

During surgery as the earlier hemostasis is achieved, the shorter time of operation, the less need for transfusion, the better is the handling of the patient and the earlier their recovery. Therefore, the shorter is the length of stay in the intensive care unit and the hospitalization, which will result in a reduced costs.

In cardiovascular surgery, especially in aortic operations, whose surgical procedure requires anticoagulation with heparin, cardiopulmonary bypass, several degrees of hypothermia, sometimes systemic circulatory arrest, among other tactics in the operative handling, all the additional resources that may help in the hemostasis are vital to improve the outcomes.

Hemostats or adhesives derived from collagen or hydrogels are products that have been developed to contain minor, less intense bleeds and act as a barrier of containment when placed on a bloody surface that in contact with the blood, would help in the formation of the clot. The sealants are basically divided into the fibrin glues (human or animal origin), products that mimic the final pathway of the coagulation cascade in the formation of the fibrin clot. Also there are the synthetic sealants (polyethylene glycol polymers) that form an adhesive over the applied site.

TDM-621 (PuraStat® component) is an absorbable, local hemostatic agent composed of nanofibers of a self-supporting polypeptide that forms a hydrogel that, when in contact with blood, allows the suture vessel wall to be optimized for hemostasis.

The hypothesis is that the use of TDM-621 may reduce bleeding and the need for blood transfusion of patients undergoing thoracic ascending aortic surgeries.

SASH Trial is a multicenter, prospective, open and randomized 1: 1 study. The aim of this study is to evaluate the effectiveness of TDM-621 on hemostasis of ascending aortic surgery. It will be performed in 5 different centers.The study will include 200 patients with ascending aortic disease according to inclusion criteria.

The protocol, informed consent form and other documents related to the study were submitted to the Ethics Committee/Institutional Review Board and was approved. The study will be carried out in accordance with the Declaration of Helsinki and Good Clinical Practices (GCP).

Statistical analysis The sample size for the study was calculated by estimating a reduction of 400 ml to 500 ml peri-operative bleeding with a standard deviation of ± 250 ml for the treated group, alpha = 5% and 80% power. To do so, it will take 99 Participants for each group, totaling 198 Participants for the study.

Categorical variables will be assessed using the chi-square test or Fisher's exact test or likelihood ratio.

The normality of the quantitative variables will be evaluated with the Shapiro-Wilks test. The parametric variables will be described with mean and standard deviation and compared with the t-Student test. Non-parametric variables will be described with median and interquartile range and compared with the Mann-Whitney test.

Values of p <0.05 will be considered significant.

Data Storage It is expected that all data entered in the eCRF will have source documentation available in the clinical center. The site must implement processes to ensure that this happens.

Quality Assurance and Data Management Data collection will be performed through an electronic CRF (eCRF). The investigator or an authorized member of the research team must sign all completed eCRFs using an electronic signature (a password will be provided by the data management center at the beginning of the study). Clinical data management will be performed according to data cleansing procedures. This is applicable for data recorded in the eCRF, as well as for data from other sources (eg laboratory tests, ECG, etc.). Proper computer editing programs will be run to verify the accuracy of the database. The researcher will be asked about incomplete, inconsistent or absent data.

The study was submitted to the Scientific and Ethics Committee of the five hospitals involved. The Managing Center, which will determine the independent randomization of the other Centers, as well as coordinate and audit the data is the Heart Institute (InCor) University of Sao Paulo General Hospital. A study-specific database will be assembled and stored on the REDCAP platform.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be over 18 years old,
2. Patient with aortic root aneurysm and / or ascending aorta, or chronic Stanford A dissections whose surgical correction is restricted to the root, ascending aorta and extending distally up to the hemiarch , including reoperations,
3. All procedures on the aortic valve and coronary ostia are allowed,
4. All patients will be clarified on the details of the study and if they agree to participate, they will sign the informed consent form.

Exclusion Criteria:

1. Patients with acute aortic dissection,
2. Patients whose correction includes total replacement of the aortic arch or distal extension to it,
3. Patients who require associated procedures on the other cardiac valves other than the aortic valve,
4. Patients who require myocardial revascularization,
5. Patients who refuse to receive blood products,
6. Patients with chronic anemia (hemoglobin less than 12g / dl for women and 13g / dl for men),
7. Platelet count less than 150,000 / mm3,
8. Coagulopathy (previous history, use of anticoagulants not reversed, prothrombin time higher than 14.8 seconds or INR (international normalized ratio) higher than 1.2), hypofibrinogenemia (fibrinogen less than or equal to 150mg / dl),
9. Patients in uninterrupted use of antiplatelet therapy (less than 7 days of operation), inhibitors of glycoproteins IIb / IIIa, as well as some supplements or vitamins (ginger, ginkgo biloba or fish oil),
10. Patients with terminal liver disease, renal dialysis and neoplasias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the total bleeding up to 48 hours of the operation. | Total blood volume measured up to 48hours after surgery.
  This evaluation will be made by measuring the wet weight of the compresses after infusion of protamine until the closure of the chest, also by measuring the volume of red cells recovered by the cell saver and through the flow of the mediastinum drain in the first 6hours, 12hours, 24hours and 48hours of the postoperative period initiated after the sternum closure.
Evaluate the number of bags of red blood cells transfused up to 48 hours of the operation. | Total amount of red cells bags up to 48hours postoperative period.
  This outcome will be evaluated by quantifying the number of bags of red blood cells needed, following the study criteria, during the operation until 48 hours after the postoperative period.

SECONDARY OUTCOMES:
To evaluate the transfusion of platelet concentrate, or cryoprecipitates or fresh frozen plasma received intraoperatively up to 48 hours after the end of the procedure. | Total number of bags of any component from intraoperative up to 48hours postoperative period.
  Number of bags transfusion of platelet concentrate,or cryoprecipitates or fresh frozen plasma, received intraoperatively up to 48 hours after the end of the procedure.
Evaluation of postoperative complications. | From the postoperative time until the date of first documented event or date of hospital discharge whichever came first up to 2 weeks.
  Surgical wound infection, mediastinitis, pulmonary infection, sepsis, low cardiac output, adult respiratory distress syndrome, acute renal failure, renal dialysis, postoperative cerebrovascular accident, convulsive crisis, delirium, deep vein thrombosis, pulmonary thromboembolism, postoperative acute myocardial infarction, atrial and ventricular arrhythmias, until the day of hospital discharge.
In hospital mortality | From the postoperative time until the date of death from any cause or date of hospital discharge whichever came first up to 2 weeks.
  In hospital mortality
Evaluation of postoperative complications. | From the postoperative time up to 72 hours and after 72 hours up to hospital discharge.
  Body temperature higher or equal 37.8 °C in the first 72 hours postoperative (with or without antibiotic therapy), temperature higher than or equal to 37.8 ° C after 72 hours postoperative (with or without antibiotic therapy).
Evaluation of postoperative complications. | From the postoperative time up to 48 hours.
  The use of vasopressors in the first 48 hours postoperatively (noradrenaline and / or vasopressin).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo R Dias, MD,PhD, Study Chair — Instituto do Coração - INCORHCFMUSP
Locations (1):
- Heart Institute (InCor) University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It is not yet decided with executive committee how and what to share IPD (individual participant data).

REFERENCES:
- [Background] Bhamidipati CM, Coselli JS, LeMaire SA. BioGlue in 2011: what is its role in cardiac surgery? J Extra Corpor Technol. 2012 Mar;44(1):P6-12. PMID 22730865
- [Background] Vyas KS, Saha SP. Comparison of hemostatic agents used in vascular surgery. Expert Opin Biol Ther. 2013 Dec;13(12):1663-72. doi: 10.1517/14712598.2013.848193. Epub 2013 Oct 22. PMID 24144261
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Management. Practice guidelines for perioperative blood management: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Management*. Anesthesiology. 2015 Feb;122(2):241-75. doi: 10.1097/ALN.0000000000000463. No abstract available. PMID 25545654
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Background] Pagano D, Milojevic M, Meesters MI, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Boer C. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):79-111. doi: 10.1093/ejcts/ezx325. No abstract available. PMID 29029100
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613
- See also: Inpatient surgery. Centers for Disease Control and Prevention; 2013. Fast Stats. — http://www.cdc.gov/nchs/fastats/inpatient-surgery.htm